CLINICAL TRIAL: NCT03044132
Title: A Prospective Trial Measuring the Clinical Outcomes for DermACELL AWM® in Chronic Wagner Grade 3/4 Diabetic Foot Ulcers
Brief Title: DermACELL AWM® in Chronic Wagner Grade 3/4 Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeNet Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-16-002
Record Dates: First submitted 2017-02-01; First posted 2017-02-06 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Diabetic Foot Ulcer; Lower Extremity Wound
Keywords: Diabetic Foot Ulcer; DFU; Lower Extremity Wound; Skin Substitute
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter post market product evaluation of study product for deep wounds of the lower extremity
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DermACELL AWM (Experimental): Human acellular dermal matrix (ADM) recovered from human donors, decellularized, provided with at least 97% DNA removal, terminally sterilized in its final package, and ready to use.
  Interventions: Other: DermACELL AWM

INTERVENTIONS:
Other: DermACELL AWM — Decellularized regenerative human tissue matrix allograft (dermis) processed using proprietary Matracell® technology

SUMMARY:
This is a prospective, multicenter, clinical research trial evaluating the clinical outcomes of DermACELL AWM in dermal regeneration.

DETAILED DESCRIPTION:
This clinical evaluation with DermACELL AWM will explore its use in the treatment of complex soft tissue defects involving muscle, fascia, tendon, or bone exposure (Wagner Classification 3 and 4).

A total of 50 subjects will be treated with DermACELL AWM in the operating room for coverage of deep soft tissue defects in the lower extremity. Subjects will then be followed in the outpatient clinic for up to 16 weeks.

The specific aim of the study is to assess the ability of the product to sustain an optimal dermal layer. The time (days) required for wound bed preparation (granular bed after placement of DermACELL AWM) and safety data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Wagner Grade 3 or 4 complex soft tissue defect that extends below subcutaneous tissue (exposed fascia, ligament, tendon, muscle, or bone)
* target wound that is either acute or chronic (nonhealing wounds greater than 4 weeks but not greater than 1 year in duration)
* target wound that is not amendable to primary closure
* target wound deemed without any residual infection (as assessed by Investigator) or is being treated upon entry into the clinical trial
* adequate perfusion to the extremity
* laboratory assessments which represent a good potential for wound healing (liver and kidney function, nutritionally stable and diabetes control)

Exclusion Criteria:

* untreated infection of soft tissue or bone
* untreated autoimmune connective tissue disorders
* body mass index (BMI) of ≥ 50
* undergoing chemotherapy/radiation therapy or taking an immunosuppressant medication
* active liver disease (e.g. hepatitis A-G),
* have undergone previous wound care therapy that included any bioengineered alternative tissue or STSG 30 days prior to enrollment
* pregnant
* enrolled in any other interventional clinical research trial
* an increase or decrease of more than 25% in wound area or volume from the Screening to Baseline visit.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Time (days) required for wound bed preparation (granular bed after placement of DermACELL AWM). | 112 Days
  Days required for granular bed formation

SECONDARY OUTCOMES:
Number of applications of study product required to achieve granulation. | 16 Weeks
Percent wound area reduction and percent complete wound closure at 16 Weeks. | 16 Weeks
The number of adverse events after DermACELL AWM application including infection, hospitalization, and reoperation. | 16 Weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Limb Preservation Platform, Fresno, California
  - Purvis Moyer Foot and Ankle Center, Rocky Mount, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cazzell S, Moyer PM, Samsell B, Dorsch K, McLean J, Moore MA. A Prospective, Multicenter, Single-Arm Clinical Trial for Treatment of Complex Diabetic Foot Ulcers with Deep Exposure Using Acellular Dermal Matrix. Adv Skin Wound Care. 2019 Sep;32(9):409-415. doi: 10.1097/01.ASW.0000569132.38449.c0. PMID 31361269